CLINICAL TRIAL: NCT05704374
Title: The Effect of Sympathetic Dysfunction on Muscle Spindle Activity in Patients With Fibromyalgia Syndrome
Brief Title: The Effect of Sympathetic Dysfunction on Muscle Spindle in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IstanbulPMRTRH-Fibromyalgia
Record Dates: First submitted 2023-01-07; First posted 2023-01-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin; Autonomic Nerve Block

STUDY DESIGN:
Who Masked: Investigator
Masking Description: In order to ensure that the researcher who took the recordings is blind, sympathetic tone measurement will be made at rest and during the sympathetic stimulation maneuver in healthy subjects 1.5 hours later, and H-reflex and T-reflex recordings will be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fibromyalgia group (Experimental): In the first phase of the experiment, the effect of sympathetic tone change on T- and H-reflexes will be evaluated.
  In the second phase of the experiment, 150 mg (single dose) of pregabalin will be given to these patients to reduce sympathetic activity and evaluate its effect on T- and H-reflexes.
  Interventions: Diagnostic Test: sympathetic stimulation maneuver (mental arithmetic test, cold pressure test); Drug: Pregabalin 150mg
- Healthy control group (Other): The effect of sympathetic tone changes on T- and H-reflexes will be evaluated in healthy cases.
  Interventions: Diagnostic Test: sympathetic stimulation maneuver (mental arithmetic test, cold pressure test)

INTERVENTIONS:
Diagnostic Test: sympathetic stimulation maneuver (mental arithmetic test, cold pressure test) — Mental arithmetic calculation and cold pressure increase sympathetic tone. For the mental arithmetic task, the subject is asked to mentally subtract a two-digit number from a four-digit number and respond within 5 seconds. This arithmetic calculation is repeated for different numbers. This test is continued for three minutes. For the cold pressure test, subjects are asked to immerse their right hand in 2-4 degrees cold water up to the elbow and hold it in the water for three minutes. The mental arithmetic task and cold stress test will be applied simultaneously.
Drug: Pregabalin 150mg — In the second phase of the experiment, 150 mg (single dose) of pregabalin will be given to FMS patients to reduce sympathetic activity and evaluate its effect on T- and H-reflexes.
  Other Names: sympathetic block
  Arms: Fibromyalgia group

SUMMARY:
This study aims to reveal whether there is an impairment in the sympathetic regulation of muscle spindle sensitivity in patients with fibromyalgia syndrome (FMS).

DETAILED DESCRIPTION:
The common muscle pain and fatigue symptoms of FMS can be explained by impaired sympathetic regulation of muscle spindle sensitivity. The aim of this study is to reveal whether there is an impairment in the sympathetic regulation of muscle spindle sensitivity in FMS patients.

Material method:

In the first stage, resting sympathetic tone measurement and resting H-reflex and T-reflex recordings will be taken in all cases. Sympathetic tone measurement will be performed and H-reflex and T-reflex recordings will be taken during and after sympathetic stimulation maneuvers (mental arithmetic calculation and cold application) in FMS patients and healthy control subjects. In the second phase, the first dose of pregabalin will be given to patients diagnosed with FMS and prescribed pregabalin. Pregabalin is known to reduce sympathetic activity in FMS. After oral administration of pregabalin, its peak plasma concentration is reached in 0.9-1.3 hours. Therefore, 1.5 hours later, sympathetic tone measurement will be made at rest and during the sympathetic stimulation maneuver, and H-reflex and T-reflex recordings will be taken. Patients in the healthy control group will not be given pregabalin.

ELIGIBILITY:
Inclusion Criteria:

For the fibromyalgia group

* Patients diagnosed with FMS based on the American college of rheumatology - 2016 criteria
* Between the ages of 20-50
* Being a woman
* Patients prescribed pregabalin for the treatment

For the Healthy Control group

* Between the ages of 20-50
* Being a woman
* Being healthy

Exclusion Criteria:

* Those with medical problems in the right upper and lower extremities (skin, neuromuscular, joint, vascular pathologies)
* Cases that cannot perform arithmetic operations
* Cold allergy
* Heart disease (arrhythmia, ischemic heart disease, heart failure)
* Hypertension
* Epilepsy

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in T-reflex amplitude after intervention | immediately after the intervention
  In order to elicit the right soleus T-reflex, a constant-intensity strike will be made on the Achilles tendon with a reflex hammer at intervals of 10-15 seconds. An accelerometer will be placed over the Achilles tendon to measure T-reflex latency and confirm that strike intensities are constant. Recordings will be taken from the right soleus muscle. T-reflex peak-to-peak amplitudes will be measured in electromyographic recordings.
Change from baseline in H-reflex amplitude after intervention | immediately after the intervention
  The right tibial nerve will be stimulated with a monopolar technique from the popliteal region to elicit the soleus H-reflex response. The stimulation electrode (cathode) will be placed on the tibial nerve in the popliteal fossa and the anode will be placed on the prepatellar region. For stimulation, a 1ms monophasic square wave pulse current will be given. Mmax will be determined firstly.The current intensity providing a 10% Mmax response will be used to test the H-reflex response. H-reflex peak-to-peak amplitude will be measured in electromyographic recordings.

SECONDARY OUTCOMES:
Heart rate variability | immediately after the intervention
  Sympathetic tone will be evaluated by measuring heart rate variability in the ECG recording taken from the DII lead.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA AYDIN, Principal Investigator — İstanbul Physical Therapy Rehabilitation Training & Research Hosptial
Locations (1):
- Tugba Aydin, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bair MJ, Krebs EE. Fibromyalgia. Ann Intern Med. 2020 Mar 3;172(5):ITC33-ITC48. doi: 10.7326/AITC202003030. PMID 32120395
- [Background] Aguilar-Ferrandiz ME, Casas-Barragan A, Tapia-Haro RM, Rus A, Molina F, Correa-Rodriguez M. Evaluation of sympathetic adrenergic branch of cutaneous neural control throughout thermography and its relationship to nitric oxide levels in patients with fibromyalgia. J Therm Biol. 2021 Jan;95:102813. doi: 10.1016/j.jtherbio.2020.102813. Epub 2020 Dec 14. PMID 33454042
- [Background] Reyes Del Paso GA, de la Coba P. Reduced activity, reactivity and functionality of the sympathetic nervous system in fibromyalgia: An electrodermal study. PLoS One. 2020 Oct 29;15(10):e0241154. doi: 10.1371/journal.pone.0241154. eCollection 2020. PMID 33119628
- [Background] Radovanovic D, Peikert K, Lindstrom M, Domellof FP. Sympathetic innervation of human muscle spindles. J Anat. 2015 Jun;226(6):542-8. doi: 10.1111/joa.12309. PMID 25994126
- [Background] Kamibayashi K, Nakazawa K, Ogata H, Obata H, Akai M, Shinohara M. Invariable H-reflex and sustained facilitation of stretch reflex with heightened sympathetic outflow. J Electromyogr Kinesiol. 2009 Dec;19(6):1053-60. doi: 10.1016/j.jelekin.2008.11.002. Epub 2008 Dec 19. PMID 19101166
- [Background] Hjortskov N, Skotte J, Hye-Knudsen C, Fallentin N. Sympathetic outflow enhances the stretch reflex response in the relaxed soleus muscle in humans. J Appl Physiol (1985). 2005 Apr;98(4):1366-70. doi: 10.1152/japplphysiol.00955.2004. Epub 2004 Nov 12. PMID 15542572
- [Background] Meeus M, Goubert D, De Backer F, Struyf F, Hermans L, Coppieters I, De Wandele I, Da Silva H, Calders P. Heart rate variability in patients with fibromyalgia and patients with chronic fatigue syndrome: a systematic review. Semin Arthritis Rheum. 2013 Oct;43(2):279-87. doi: 10.1016/j.semarthrit.2013.03.004. Epub 2013 Jul 6. PMID 23838093
- [Background] Light KC, Bragdon EE, Grewen KM, Brownley KA, Girdler SS, Maixner W. Adrenergic dysregulation and pain with and without acute beta-blockade in women with fibromyalgia and temporomandibular disorder. J Pain. 2009 May;10(5):542-52. doi: 10.1016/j.jpain.2008.12.006. PMID 19411061
- [Background] White AT, Light KC, Bateman L, Hughen RW, Vanhaitsma TA, Light AR. Effect of Pregabalin on Cardiovascular Responses to Exercise and Postexercise Pain and Fatigue in Fibromyalgia: A Randomized, Double-Blind, Crossover Pilot Study. Pain Res Treat. 2015;2015:136409. doi: 10.1155/2015/136409. Epub 2015 Dec 29. PMID 27026828
- [Background] Bockbrader HN, Radulovic LL, Posvar EL, Strand JC, Alvey CW, Busch JA, Randinitis EJ, Corrigan BW, Haig GM, Boyd RA, Wesche DL. Clinical pharmacokinetics of pregabalin in healthy volunteers. J Clin Pharmacol. 2010 Aug;50(8):941-50. doi: 10.1177/0091270009352087. Epub 2010 Feb 10. PMID 20147618